CLINICAL TRIAL: NCT06472843
Title: Tailoring Upper Limb Exercise Advice for People With Parkinson Disease
Acronym: ICEBERG
Status: Not yet recruiting | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Daryl Wile, Clinical Assistant Professor, University of British Columbia Southern Medical Program, University of British Columbia
Other Study IDs: 001
Record Dates: First submitted 2024-04-23; First posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Parkinson Disease; Upper Limb; Aerobic Exercise
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Interval: Participants in the interval condition will begin with a gradual one minute warm up effort with a ramp in the resistance gradually increasing from 0 watts to 60% of their peak power output (Wpeak) over 1 minute. They will then perform five sets of high intensity intervals with rest between these efforts. The intervals will be at 100% Wpeak for 15 seconds followed by 60% Wpeak for 45 seconds. During the work intervals participants will be encouraged to apply the highest cadence they can produce for the 15 second interval and resume a freely chosen cadence in the rest periods. After five interval repetitions (5 minutes) they will gradually warm-down from 60% Wpeak to 0 watts over 1 minute.
  Interventions: Behavioral: Exercise Intervention
- Steady State: Participants in the steady state condition will begin the intervention with a gradual one minute warm up effort with a ramp in the resistance gradually increasing from 0 watts to 70% of their Wpeak over 1 minute. They will then continue at this resistance level at a freely chosen cadence for 5 minutes, after which they will gradually warm-down to 0 watts over 1 minute.
  Interventions: Behavioral: Exercise Intervention

INTERVENTIONS:
Behavioral: Exercise Intervention — The exercise session is a fitness test using a hand bike, and you will be randomly assigned to one of two exercise sessions. The fitness test and exercise sessions are short (less than 10 minutes).

SUMMARY:
The investigators will explore the impact of hand cycling, on hand function in people with Parkinson's Disease (PD). The study will compare the effects of two different hand cycling approaches-steady-state and interval efforts-on improving hand dexterity in people with PD. Conducted as a clinical trial, it aims to understand if a single session of hand cycling can temporarily enhance hand function and if the nature of the exercise influences the benefit.

DETAILED DESCRIPTION:
The purpose of this study is to examine the effects of hand cycling, an upper limb aerobic exercise, on hand function in individuals with Parkinson's Disease (PD).

Parkinson's Disease affects motor skills, including hand dexterity, which can impede daily activities. While aerobic exercise is known to have benefits for people with PD, the specific impact of upper limb exercises like hand cycling on hand function is less studied. Previous research suggests aerobic exercises can improve symptoms and motor function in PD. This study aims to fill the gap in understanding how hand cycling affects hand dexterity in PD. There is no placebo involved in this study as it compares two active intervention types: steady-state and high-intensity interval hand cycling.

This is a block randomized parallel group clinical trial involving a single session of exercise intervention. Participants will be randomly assigned to one of two groups: steady-state or high-intensity interval hand cycling. The study includes baseline assessments, the exercise intervention, and post-intervention assessments to evaluate changes in hand function.

The primary endpoint is the time to complete the 9-hole pegboard test with the clinically more affected hand. Secondary endpoints include changes in motor examination scores, finger tapping speed, and subjective measures of exercise perception. Analysis of covariance will be used to compare the primary outcome between groups, accounting for baseline performance and clinical characteristics. The planned sample size is 20 people with PD, aiming to capture varied clinical expressions of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 19 with a clinical diagnosis of PD.

Exclusion Criteria:

* Medical contraindication to aerobic exercise, such as unstable cardiovascular disease, or physical disability that precludes arm exercise.
* Individuals will be excluded if, upon screening with the Canadian Society for Exercise Physiology (CSEP) Get Active Questionnaire and International Physical Activity Questionnaire Short Form (IPAQ-SF) a need for further evaluation before exercise is identified

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with Parkinson Disease that are medically fit to perform a brief session of aerobic exercise.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
9-hole pegboard test | Through study completion, an average of 9 months
  Time to complete the 9-hole pegboard test with the clinically more affected hand.

SECONDARY OUTCOMES:
Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS III) score | Through study completion, an average of 9 months
  Motor subscale of the movement disorders society revised unified Parkinson Disease Rating Scale
Finger tapping speed | Through study completion, an average of 9 months
  Number of alternate finger taps completed in a 30 second period in each hand
Perceived exertion | Through study completion, an average of 9 months
  Borg Category Ratio (CR)10 rating of perceived exertion (RPE) scale
Positive Affect | Through study completion, an average of 9 months
  Self-reported positive-activated affect (PAA) two-dimensional likert scale
Enjoyment | Through study completion, an average of 9 months
  Exercise Enjoyment (Likert scale)

IPD SHARING:
Plan to Share IPD: Undecided